CLINICAL TRIAL: NCT02064348
Title: A Thorough QTc Evaluation of the Effect of Semaglutide on Cardiac Repolarisation in Healthy Subjects: A Randomised, Double-Blind,Placebo-Controlled, Three-Arm Parallel Trial With a Nested Cross-Over Design for Positive Control With Moxifloxacin Administration
Brief Title: A Thorough QTc Evaluation of the Effect of Semaglutide on Cardiac Repolarisation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3652; 2012-005073-31 (EudraCT Number); U1111-1136-6455 (Other: WHO)
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: semaglutide + moxifloxacin placebo (Experimental): Subjects will receive a single dose of moxifloxacin placebo both before the start of semaglutide treatment and at the end of the semaglutide treatment.
  Interventions: Drug: semaglutide; Drug: placebo
- Arm 2A: (Active Comparator): Semaglutide placebo + moxifloxacin/moxifloxacin placebo:
  Subjects will receive moxifloxacin before the start of semaglutide placebo treatment and moxifloxacin placebo at the end of the semaglutide placebo treatment.
  Interventions: Drug: placebo; Drug: moxifloxacin
- Arm 2B: (Experimental): Semaglutide placebo + moxifloxacin placebo/moxifloxacin:
  Subjects will receive moxifloxacin placebo before the start of semaglutide placebo treatment and moxifloxacin at the end of the semaglutide placebo treatment.
  Interventions: Drug: placebo; Drug: moxifloxacin

INTERVENTIONS:
Drug: semaglutide — Solution for subcutaneous (s.c., under the skin) injection. Dose escalation to 1.5 mg.
  Arms: Arm 1: semaglutide + moxifloxacin placebo
Drug: placebo — Solution for s.c. injection or tablets for oral administration
Drug: moxifloxacin — Tablets for oral administration
  Arms: Arm 2A:; Arm 2B:

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to evaluate the effect of semaglutide on cardiac repolarisation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index): 20-30 kg/m^2
* Body weight: 60-110 kg
* Normal ECG (electrocardiogram)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method. Women of child-bearing potential must use an effective method of birth control for the duration of the trial and for 5 weeks following the last dose of semaglutide. Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices), or sexual abstinence or vasectomised partner
* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ
* History of seizures, epilepsy, syncope, cardiac arrest, cardiac arrhythmia or Torsades de Pointes, A-V (Atrioventricular) block or structural heart disease
* Family history of long QT (Interval in the ECG: from the start of the QRS complex to the end) syndrome (either objectively diagnosed or suggested by sudden death due to cardiac causes before the age of 50 of a 1st degree relative)
* Family history of sudden cardiac death before the age of 50 of a 1st degree relative
* Use of prescription or non-prescription systemic or topical medicinal products (except routine vitamins, acetylsalicylic acid, paracetamol and contraceptives) within 3 weeks (or within 5 halflives of the medicinal product, whichever is longest) prior to the first dosing of semaglutide
* Smoking, drug or alcohol abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2015-04-23 (Actual); Study Completion 2015-04-23 (Actual)

PRIMARY OUTCOMES:
QTcI, (Individual heart rate corrected QT (Interval in the ECG: from the start of the QRS complex to the end) interval) based on ECG recordings obtained at 11 time points | 0-48 hours after the fourth dose of semaglutide/semaglutide placebo at the 1.5 mg dose level

SECONDARY OUTCOMES:
QTcI, based on ECG (electrocardiogram) recordings obtained at 2 out of 8 time points | 0-24 hours after a single dose of moxifloxacin/moxifloxacin placebo

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] Demmel V, Sandberg-Schaal A, Jacobsen JB, Golor G, Pettersson J, Flint A. No QTc Prolongation with Semaglutide: A Thorough QT Study in Healthy Subjects. Diabetes Ther. 2018 Aug;9(4):1441-1456. doi: 10.1007/s13300-018-0442-0. Epub 2018 May 24. PMID 29799100
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com